CLINICAL TRIAL: NCT05870605
Title: Drug Utilisation Study of Intuniv® (Guanfacine Extended Release) in European Countries
Brief Title: Drug Use Study With Intuniv® in European Countries
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP503-802; EUPAS18739 (Other: EU PAS Registry); EUPAS18735 (Other: EU PAS Registry)
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Drug Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Database Survey: All prescriptions for Intuniv available in the database in Denmark, Germany, Norway, Spain, Sweden, and the United Kingdom will be analyzed.
  Interventions: Other: No Intervention
- Physician Survey: The physicians will collect participant records of those who have been prescribed Intuniv® at least once during the study period of 4 years. This will be done in Belgium, Finland, Ireland, and the Netherlands.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observational study utilizing historical de-identified patient level data; therefore no intervention is given.

SUMMARY:
This study will evaluate and characterize people who are taking Intuniv, analyze prescribing behaviors of physicians, and determine whether Intuniv was correctly prescribed in Belgium, Denmark, Finland, Germany, Ireland, Netherlands, Norway, Spain, Sweden, and the United Kingdom.

DETAILED DESCRIPTION:
The study aims to characterize participants who are prescribed Intuniv® and describe prescribing patterns of Intuniv® among physicians in European countries.

This study will collect data from the following sources:

* Physician Survey: de-identified patient data provided by representative physicians in Belgium, Finland, Ireland, and the Netherlands, with a goal of data from up to 100 participants per survey wave.
* Database Survey: longitudinal patient-level prescription database in all other countries with data on approximately 5000 participants.

In the database study, actual prescription data are collected from electronic medical records and national registries. A prescriber survey will be conducted to evaluate health care professionals (HCPs) real-life practice. It will include data collection from the prescriber's (physician's) files and a web questionnaire, including de-identified data from up to 100 participants per survey wave.

ELIGIBILITY:
Inclusion Criteria:

* Prescribers of Intuniv®, i.e. physicians who know and have prescribed the drug at least once during the previous 12 months (or, for the first report, since country specific launch) (paediatricians, psychiatrists, neurologists and GPs).
* Participants who have been prescribed Intuniv® at least once during the reporting period.

Exclusion Criteria:

• Physicians who do not treat participants or who may have a conflict of interest (i.e. physicians employed by regulatory bodies or pharmaceutical industries).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prescribers of Intuniv® in the European countries.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Stratified by Prescriber Information Based on Physician Survey | Up to 4 years
  Participants will be stratified based on prescriber information which include demographics, specialty, and setting of prescriber.
Number of Participants Categorised Based on Their Demographic Characteristics | Up to 4 years
  The demographic characteristics will include age and gender.
Number of Participants with Co-morbidities | Up to 4 years
Number of Participants Based on Indication of Use of Prescribed Intuniv® | Up to 4 years
  Indication of use (diagnosis) will be assessed as per World Health Organization (WHO) 10th International Statistical Classification of Diseases and Related Health Problems (ICD) classification.
Number of Participants With ADHD Categorised Based on Different Patterns of Intuniv® Use | Up to 4 years
  Patterns of drug use include first time users, repeat users, participants who discontinued the ADHD therapy, participants with switches in treatment (both from Intuniv® to other ADHD medications and other ADHD medications to Intuniv®), and participants with dosing/overdose (defined as daily dose of >7 mg or of >4mg in participants ≤12 years of age).
Number of Participants Using Intuniv® as Second Line Treatment After Psychostimulant Prescription at any Time Prior to the Participant's First Prescription of Intuniv® | Up to 4 years

SECONDARY OUTCOMES:
Number of Physician Visits During the First Year of Therapy | Up to 4 years
Frequency of Weight Monitoring of Participants by Physician | Up to 4 years
  Frequency of weight monitoring of participants by physician will be reported.
Frequency of Blood Pressure Monitoring of Participants by Physician | Up to 4 years
  Frequency of blood pressure monitoring of participants by physician will be reported.
Frequency of Heart Rate Monitoring of Participants by Physician | Up to 4 years
  Frequency of heart rate monitoring of participants by physician will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Real World Insights EMEA IQVIA Commercial GmbH & Co. OHG, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/f02c19325d0b4658?idFilter=%5B%22SHP503-802%22%5D